CLINICAL TRIAL: NCT02458274
Title: Circulating and Pulmonary Microparticles for Early Diagnosis of Bronchiolitis Obliterans Syndrome After Lung Transplantation
Brief Title: Microparticles and Bronchiolitis Obliterans Syndrome
Acronym: MIBO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5254
Record Dates: First submitted 2015-04-14; First posted 2015-06-01 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Broncho-alveolar lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient without bronchiolitis obliterans syndrome: Lung transplanted patient without bronchiolitis obliterans syndrome
  Interventions: Other: Dosage of Microparticles (MPs) in broncho-alveolar lavage fluid (BALF)
- Patient with bronchiolitis obliterans syndrome: Patient with bronchiolitis obliterans syndrome three years after lung transplantation.
  Interventions: Other: Dosage of Microparticles (MPs) in broncho-alveolar lavage fluid (BALF)

INTERVENTIONS:
Other: Dosage of Microparticles (MPs) in broncho-alveolar lavage fluid (BALF)

SUMMARY:
The main long-term complication of lung transplantation is chronic lung allograft dysfunction (CLAD). Bronchiolitis obliterans syndrome (BOS) is the most frequent presentation of CLAD. BOS leads to a progressive loss of lung allograft function, with recurrence of dyspnea and airflow limitation. In some advanced cases, patients need a lung re transplantation. The mechanisms of BOS are not completely elucidated, and there are no early markers or specific treatment available for this condition.

Microparticles (MPs) are submicron plasma membrane fragments released into the vascular compartment or the pericellular space in response to cell activation, injury or apoptosis. Broncho alveolar and circulating MPs may reflect cellular insults of the lung allografts. Therefore, MPs could be viewed either as biomarkers or as effectors of the chronic inflammatory or procoagulant processes leading to bronchiolitis obliterans syndrome.

The investigators plan to include 60 patients before lung transplantation at our centre in Strasbourg (France). Follow-up will be requested at the base of usual care (spirometry, blood sampling, bronchoscopy with broncho-alveolar lavage [BAL]). The investigators will measure at one month, one, two and three year post transplantation, the total concentration of MPs in plasma and BAL and characterize their phenotype.

The investigators objective is to demonstrate correlation between total MPs concentration in broncho-alveolar lavage fluid (BALF) and the occurrence of bronchiolitis obliterans syndrome at three years post lung transplantation.

ELIGIBILITY:
Inclusion criteria:

* Every adult (>18 years) patient on lung transplant waiting list
* Patients who give a written informed consent
* Patients affiliated to a social security regimen

Exclusion criteria:

* Patients on lung transplant waiting list for BOS
* Patients who cannot sign an informed consent form (emergency situation, patient with understanding difficulties…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with a lung transplantation will be included in one center (Strasbourg) 30 -40 lung transplantations are performed each year in our centre, with a survival rate of 80% at three year post transplantation. Approx. 30% patients will develop BOS at three year post transplantation. So we expect at three year post transplantation 15 patients with BOS and 37 patients without BOS (52 patients alive at three years post transplantation).
  Consequently, the total duration of the study will be five years (two years for inclusion and three years of follow-up)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2020-05 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Correlation between total concentration of MPs in broncho-alveolar lavage fluid (BALF) and occurrence of bronchiolitis obliterans syndrome at three year post lung transplantation | Lung transplanted patients will be followed up with usual care. Spirometry and bronchoscopy with BALF at three years after transplantation will be used in the present study.
  We will measure at three years post transplantation, the total concentration of MPs in plasma and BAL and characterize their phenotype Bronchiolitis Obliterans Syndrome (BOS) will be graded according to guidelines of the the International Society for Heart and Lung transplantation. Percentage of decrease of lung function based on actual FEV1 compared to the average of the two best FEV1, distant for three week, post lung transplantation.
  BOS 0 : FEV1 > 90% BOS 0-p : 90 >FEV1 > 81% BOS 1 : 80 >FEV1 > 66% BOS 0-p : 65 >FEV1 > 51% BOS 0-p : FEV1 < 50% If BOS is present, we usually do CT-scan and bronchoscopy with BALF to confirm BO and eliminate alternative diagnosis.

SECONDARY OUTCOMES:
Total concentration MPs and characterization of cellular origin of MPs in BALF and in plasma of patients at three year post lung transplantation. | Lung transplanted patients will have spirometry and bronchoscopy with BALF at three years after transplantation as it's usually done for each lung transplanted.
  MPs expose to the surface phosphatidylserine (PhtdSer), tissue factor and membrane antigens from the parental cells.
  MPs collected from plasma and BALF will have differential centrifugation and concentrations of MPs will be measured using original functional multiwell assays.
  MPs will be captured onto annexin-5 (total MPs) or onto specific antibodies directed against membrane antigens borne by MPs and testifying their cell origin (CD104, CD66b, CD62E, CD62P, CD35, E105, CD14, CD3, CD20).

CONTACTS AND LOCATIONS:
Overall Officials: Leclercq Alexandre, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- CHU Strasbourg, Strasbourg, France